CLINICAL TRIAL: NCT07198932
Title: Effectiveness and Safety of Cofrogliptin and Linagliptin as add-on Therapy to Insulin in Chinese Adults With Type 2 Diabetes Mellitus: a Multicenter, Prospective Real-world Study (COLOR-REAL)
Brief Title: Cofrogliptin and Linagliptin as add-on Therapy to Insulin in Type 2 Diabetes
Acronym: COLOR-REAL
Status: Not yet recruiting | Type: Observational
Sponsor: Yanbing Li (Other)
Responsible Party: Sponsor-Investigator, Yanbing Li, First Affiliated Hospital, Sun Yat-Sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: IIT-2025-340
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: real-world study; cofrogliptin; DPP-4i; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cofrogliptin cohort
  Interventions: Drug: Cofrogliptin add to insulin
- Linagliptin cohort
  Interventions: Drug: Linagliptin add to insulin

INTERVENTIONS:
Drug: Cofrogliptin add to insulin — Patients will be treated with commercially available cofrogliptin according to routine clinical practice at the discretion of the treating physician.
  Groups: Cofrogliptin cohort
Drug: Linagliptin add to insulin — Patients will be treated with commercially available linagliptin according to routine clinical practice at the discretion of the treating physician.
  Groups: Linagliptin cohort

SUMMARY:
This study is a multicenter, prospective, non-interventional real-world study to evaluate the clinical outcomes of biweekly cofrogliptin versus daily linagliptin as an add-on therapy in Chinese adult T2D patients.

DETAILED DESCRIPTION:
About 43 hospitals from different parts of China will take part in this study. Patients aged ≥18 years who have been previously treated with a stable dose of insulin and no more than three classes of oral antidiabetic drugs (OADs) for at least 12 weeks without adequate glycemic control will be enrolled and assigned to either cofrogliptin once every 2 weeks cohort or linagliptin once-daily cohort based on the prescription. Initiation of cofrogliptin or linagliptin treatment was at the treating physician's discretion.

Enrolled participants will undergo routine follow-up for up to 24 weeks. During the follow-up period, data will be collected from face-to-face participant-investigator visits at the beginning of the study (0 weeks, visit 1), early stage (4 weeks, visit 2), mid-stage (12 weeks, visit 3) and at the end of the study (24 weeks, visit 4). Data sources include patient medical records, diaries, self-monitoring of blood glucose (SMBG), and questionnaires. No additional diagnostics, monitoring procedures, or interventions outside of usual clinical practice will be applied to the participants. The project will probably last for about 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form.
2. Aged ≥18 years.
3. Diagnosed with type 2 diabetes mellitus (meeting the 1999 WHO diagnostic criteria).
4. Recently tested HbA1c 7%-9% and FPG ≤11 mmol/L, with stable treatment using insulin ± OADs for at least 12 weeks prior to enrollment. Insulin regimens are limited to: basal insulin once daily or once weekly, premixed insulin once or twice daily, or IDegAsp once or twice daily. OAD classes are limited to metformin, SGLT2 inhibitors, and α-glucosidase inhibitors and with no more than three agents in total.
5. Willing to start or have already initiated cofrogliptin or linagliptin treatment (at the physician's discretion in accordance with clinical practice). The treatment decision is independent of study enrollment, must be made before signing the informed consent, and cofrogliptin or linagliptin initiation must occur either within 2 weeks before or within 2 weeks after signing the informed consent.

Exclusion Criteria:

1. Allergic to the study drug.
2. Diagnosed with type 1 diabetes.
3. Unable to comply with study-specific procedures.
4. Current or planned pregnant, or currently breastfeeding.
5. With any other situation judged by the investigator, that is unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world adult population with type 2 diabetes in China.
Sampling Method: Non-Probability Sample
Enrollment: 594 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to 24 weeks

SECONDARY OUTCOMES:
Change in HbA1c | from baseline to 12 weeks
Reaching of HbA1c target (defined as HbA1c less than 7%) | at 24 weeks
  Percentage point
Change in FPG | from baseline to 24 weeks
  mmol/L
Change in PPG | from baseline to 24 weeks
  mmol/L
Change in fasting C peptide | from baseline to 24 weeks
  ng/mL
Change in body weight | from baseline to 24 weeks
  Kg
Change in insulin dose | from baseline to 24 weeks
  units/day
Overall safety, consisting of adverse events (AEs), serious adverse events (SAEs), adverse events of special interest | from baseline to 24 weeks

OTHER OUTCOMES:
Diabetes Treatment Satisfaction Questionnaire status (DTSQs) | at baseline, 12 weeks and 24 weeks
  questionnaire scores
Short-Form 36 Health Survey (SF-36) | at baseline, 12 weeks and 24 weeks
  questionnaire scores
Drug adherence | at 24 weeks
  measured by pill counts
Drug persistence | at 24 weeks
  defined as the proportion of patients who continued to use their index medications

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing
  - the First Medical Center of Chinese PLA General Hospital, Beijing
  - Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Xi'an International Medical Center Hospital, Xi'an